CLINICAL TRIAL: NCT05108883
Title: IDEntifying pAtients With Suspicion of Infection in the ED Who Have Low Disease Severity Using Midregional Proadrenomedullin (MR-proADM) - Pivotal Study
Brief Title: Risk Stratification Using Midregional Proadrenomedullin in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IDEAL+ Study
Record Dates: First submitted 2021-10-18; First posted 2021-11-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Patients Presenting With Suspicion of Infection to the ED

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care arm (No Intervention): decision whether a patient will be hospitalized or be treated as out-patient is based on routine clinical assessment and usual protocols
- MR-proADM guided arm (Experimental): decision whether a patient will be hospitalized or be treated as out-patient is based on routine clinical assessment, usual protocols and MR-proADM levels
  Interventions: Device: MR-proADM KRYPTOR

INTERVENTIONS:
Device: MR-proADM KRYPTOR — MR-proADM ≤ 0.87 nmol/L together with routine clinical evaluation identifies patients with low disease severity who do not need to be hospitalized
  Arms: MR-proADM guided arm

SUMMARY:
Emergency departments (ED) are becoming increasingly over-crowded, with patients facing prolonged waiting times. Therefore, a safe and rapid assessment that identifies patients with low severity that could be treated as outpatients is essential for improving the workflow within the ED.

The rationale of this IDEAL+ study is to safely decrease the number of hospital admissions through identification of low risk patients with the biomarker MR-proADM. This will has already been tested in the IDEAL - pilot study and results should be confirmed with this IDEAL+ study.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients presenting to the ED with suspicion of infection
2. Age ≥18 years
3. Written Informed Consent obtained

Exclusion Criteria:

1. Patients with SARS-COV-2 infection
2. Recent major trauma or surgery
3. End stage renal failure requiring dialysis
4. Terminal disease and/or very severe medical co-morbidity where death has to be expected in the next 6 months, e.g. due to malignancy, cardiac, renal or hepatic failure
5. Patients whose source of infection always requires hospital admission or never requires hospital admission.
6. Patients who cannot be discharged for other than medical reasons
7. Patient participates in any other interventional clinical trial
8. Patients with active abusive drug use
9. Pregnant or lactating women
10. Patients who are institutionalized by official or judicial order
11. Dependents of the sponsor, the CRO, the study site or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Number of out-patients re-presenting to the ED | 5 days
  Number of out-patients re-presenting to the ED

CONTACTS AND LOCATIONS:
Locations (9):
- Hôpital Pitié-Salpêtrière, AP-HP.Sorbonne Université, Paris, France
- Italy (2):
  - Policlinico Tor Vergata, Roma
  - Hospital Santa Maria della Misericordia, Udine
- Spain (4):
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Hospital Clinic, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen de la Macarena, Seville
- United Kingdom (2):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - University Hospital Southampton NHS Foundation Trust, Southampton